CLINICAL TRIAL: NCT01321918
Title: Register and DNA Bank of Adult Extra-hospital Sudden Death
Brief Title: Register and DNA Bank of Adult Extra-hospital Sudden Death (Protocol FASTER)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Nantes University Hospital (Other)
Responsible Party: Anne OMNES, Nantes University Hospital
Masking: None
Other Study IDs: 06/6-A; 2006-A00544-47 (Other: AFSSAPS)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Extra-hospital Sudden Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case subjects (Other)
  Interventions: Other: Case Controls
- Control subjects (Other)
  Interventions: Other: Control subjects

INTERVENTIONS:
Other: Case Controls — A blood sample of 10 ml (2 x 5 ml) on two EDTA tubes will be realised on a route of vascular development place in the context of medical practice.Clinical data will be indicated in the CRF and the computerized database. In the event an eligible patient has not been included during his support by an emergency ambulance service but, after successful resuscitation, he has been hospitalised in a cardiology department, its inclusion may be realised during the hospitalization by a physician investigator of the study. A blood sample of 10 ml of 2 EDTA tubes will be realised on a route of vascular development in the context of routine care.
  Arms: Case subjects
Other: Control subjects — A blood sample of 10 ml (2 x 5 ml) on two EDTA tubes will be realised and clinical data will be indicated in the CRF and the computerized database.
  Arms: Control subjects

SUMMARY:
The main objective of this study is the formation of a DNA bank to realise a case-control genetic study designed to identify sequence variations in DNA that predispose to sudden cardiac death in adults.

The secondary objective of this study is the creation of a register for epidemiological surveillance of adult extra-hospital sudden death.

ELIGIBILITY:
INCLUSION CRITERIA :

* Inclusion criteria for register :
* Adults ≥ 18 years of age.
* Persons who experienced sudden death defined as follows :cardiovascular arrest of non traumatic origin that occurred unexpectedly within an hour after the start of any prodromes.
* Patients not hospitalized at the time of sudden death.
* Inclusion criteria for DNA bank :
* Case subjects :
* Adults ≥ 18 years of age.
* Persons who experienced sudden death defined as follows :cardiovascular arrest of non traumatic origin that occurred unexpectedly within an hour after the start of any prodromes.
* Patients not hospitalized at the time of sudden death.
* Patients supported clinically by an emergency ambulance service.
* Control subjects :
* Adults ≥ 18 years of age.
* Adults hospitalized in an cardiac intensive care unit.

EXCLUSION CRITERIA :

* Exclusion criteria for register :
* Violent death : criminal, suicidal or accidental.
* Exclusion criteria for DNA bank :
* Case subjects :
* Violent death : criminal, suicidal or accidental.
* Identified cause of death extra-cardiac : neurological cause, hypoxia, pulmonary embolism, aortic rupture or other identified extra-cardiac cause.
* In accordance with Articles L1221-5 L1221-L1221-8 and 8-1 of the Code of Public Health, the categories of persons are excluded from research due to the fact that it can be achieved with an efficiency comparable over another class of people :
* Adult subject to legal protection measure,
* Pregnant woman,
* Parturient,
* Breastfeeding mother,
* Person deprived of liberty,
* Person hospitalised without his consent,
* Person admitted to a medical or socially facility.
* Control subjects :
* History of sudden death,
* Documented history of ventricular fibrillation,
* History of sustained ventricular tachycardia (lasting longer than 30 seconds) documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Identification of variants in DNA
  The primary endpoint is the identification of variants (polymorphisms and / or mutations) in DNA significantly associated with risk of extra-hospital sudden death in adults. Study populations are : (i) the entire population of case subjects included in the DNA bank (ii) two subpopulations at high risk of sudden death : patients with a history of myocardial infarction and patients with LVEF < 30 %. The variable analyzed is the nucleotide sequence of DNA in populations of case and control subjects.

SECONDARY OUTCOMES:
Annual incidence of extra-hospital sudden death in adults
  The annual incidence of extra-hospital sudden death in adults. The variable analyzed is the number of incident cases per year of extra-hospital sudden death in adults.
Annual mortality related to extra-hospital sudden death in adults
  The annual mortality related to extra-hospital sudden death in adults. The variable analyzed is the number of annual deaths due to sudden death in adults.
Characterization of victims of extra-hospital sudden death in adults
  The characterization of victims of extra-hospital sudden death in adults, their medical care in emergency and their future from D0 to D28. Variables analyzed are clinical data are collected in case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PROBST, Profesor, Principal Investigator — Nantes University Hospital; Jean-Luc CHASSEVENT, Doctor, Study Chair — University Hospital, Angers; Nicolas HOURDIN, Doctor, Study Chair — CH de Châteaubriant; Yves-Marie PLUCHON, Doctor, Study Chair — CH de la Roche-sur-Yon; Christophe SAVIO, Doctor, Study Chair — CH du Mans; Jean-Pierre AUFFRAY, Profesor, Study Chair — CHU de Marseille; Christian HAMON, Doctor, Study Chair — CH de Saint-Brieuc; Christophe BERRANGER, Profesor, Study Chair — CH de Saint-Nazaire; Jean-Louis DUCASSE, Doctor, Study Chair — University Hospital, Toulouse; BOULANGER, Doctor, Study Chair — CH de Vannes
Locations (1):
- Nantes University Hospital, Nantes, France